CLINICAL TRIAL: NCT05327803
Title: A Phase 2/3, Randomized, Double-blind, Placebo-controlled, Multicenter, Prospective Study to Assess the Efficacy, Safety, and Pharmacokinetics of Orally Administered Epetraborole in Patients With Treatment-refractory Mycobacterium Avium Complex Lung Disease
Brief Title: Study of Epetraborole in Patients With Treatment-refractory MAC Lung Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: EBO-301 truncated Phase 3 study (n=97) misses primary endpoint; results unable to confirm clinical efficacy observed in Phase 2 study.
Sponsor: AN2 Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EBO-301
Record Dates: First submitted 2022-03-24; First posted 2022-04-14 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-08

CONDITIONS: MAC Lung Disease; Treatment Refractory MAC Lung Disease
Keywords: NTM; Respiratory Infection; antimycobacterial activity; antimycobacterial agent; antimycobacterial therapy; MAC infections; MAC lung disease; MAC lung infection; MAC pulmonary infection; Mycobacteria; mycobacterial disease; mycobacterium; Mycobacterium Avium Complex; Mycobacterium Avium Complex Infections; Mycobacterium avium complex lung disease; Mycobacterium Infections; Nontuberculous; Nontuberculous mycobacteria / mycobacterial / mycobacterium; Non-tuberculous mycobacteria disease; Non-tuberculous mycobacterial (NTM) infections; Nontuberculous mycobacterial lung disease; Non-tuberculous mycobacterial lung disease; Nontuberculous mycobacterial pulmonary disease; NTM infection; NTM lung disease; NTM Pulmonary Disease; NTM lung infection; Pulmonary MAC disease; Pulmonary MAC lung disease; Pulmonary Mycobacterium Avium Complex disease; Treatment refractory MAC lung disease; Treatment refractory mycobacterial lung disease; Treatment refractory NTM lung disease; Treatment refractory NTM lung infection; Treatment refractory NTM pulmonary disease
MeSH Terms: conditions — Respiratory Tract Infections; Mycobacterium Infections; Mycobacterium avium-intracellulare Infection; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- epetraborole + OBR (Experimental): epetraborole + Optimized Background Regimen
  Interventions: Drug: Epetraborole
- placebo + OBR (Placebo Comparator): Placebo + Optimized Background Regimen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epetraborole — 500 mg taken orally QD
  Other Names: AN2-501971
  Arms: epetraborole + OBR
Drug: Placebo — Placebo taken orally QD
  Arms: placebo + OBR

SUMMARY:
This is a pivotal Phase 2/3, double-blind, placebo-controlled study of epetraborole + OBR (Optimized Background Regimen) versus placebo + OBR in patients with treatment-refractory MAC lung disease. This study will enroll adult patients with treatment-refractory MAC lung disease who meet all eligibility criteria (including clinical, radiographic, and microbiological criteria).

DETAILED DESCRIPTION:
In the Phase 2 part of the study, approximately 80 patients will be randomized in a 1:1 ratio (40 patients receiving active epetraborole tablets and 40 patients receiving matching placebo tablets). The Phase 2 part of the study includes a blinded psychometric analysis plan to assess the psychometric properties of a novel PRO instrument. In addition, symptom-based clinical responses will be assessed using blinded data, to inform the measurement of clinical response in the Phase 3 part of the study.

The Phase 3 part of the study will test the superiority of epetraborole + OBR compared to placebo + OBR. In this part of the study, approximately 234 patients are planned to be randomized in a 2:1 ratio (156 patients receiving active epetraborole tablets and 78 patients receiving matching placebo tablets). The current symptom-based clinical response definition (using the novel PRO) in Phase 3 is a placeholder to be verified after Phase 2 analyses based on data through Month 6. In addition, the Sponsor will determine if the sample size for Phase 3 should be adjusted and will verify the Phase 3 epetraborole dosage regimen based on the observed plasma epetraborole exposure.

Phase 3 data analyses will include a review of patient-reported outcomes, microbiological, safety, and PK data collected at multiple time points through Month 6. Patients in Phase 3 will continue double-blinded study drug for 12 months after the first negative MAC culture that defines sputum culture conversion; study drug will be discontinued in patients who remain MAC culture positive despite 6 months of therapy with study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who are 18 years of age or older.
2. Willing and able to provide written informed consent.
3. Patients with a diagnosis of treatment-refractory MAC lung disease consisting of all of the following (a) Microbiological, (b) Clinical, and (c) Radiographic criteria:

   1. Microbiological criteria:

      * One Pre-Study MAC-positive respiratory specimen. Documentation of a MAC positive specimen collected per standard of care within 6 months prior to signing the informed consent form (ICF).
      * One Screening MAC-positive expectorated or induced sputum sample.
   2. Clinical criteria: At least 2 of the following patient-reported clinical symptoms:

      * Cough with sputum production
      * Cough without sputum
      * Chest congestion
      * Hemoptysis
      * Dyspnea
      * Fatigue
      * Night sweats or unusual sweating
   3. Radiographic criteria: Non contrast Chest CT scan within 6 months prior to signing the ICF with abnormalities consistent with MAC lung disease.
   4. OBR criteria: An OBR is a combination regimen that consists of ≥2 antimycobacterial agents. The patient-specific OBR must be administered for a minimum duration of 6 consecutive months that is either ongoing at the time of Screening or was stopped or paused no more than 12 months before screening. The OBR regimen administered during Screening must be continued after randomization.
4. Patients who are willing to comply with all the study activities and procedures throughout the duration of the study and comply with all planned study visits and study procedures from Screening through the LFU Visit.
5. All patients must agree to use an effective method of birth control.
6. Patients expected to survive with continued antimycobacterial therapy and appropriate supportive care from Screening through the LFU Visit, in the judgment of the Investigator.

Exclusion Criteria:

1. Patients with a presence of any suspected or confirmed disease or condition at Screening or the time of randomization that, in the opinion of the Investigator, may confound the assessment of symptom-based clinical response.
2. Patients with active pulmonary malignancy or any malignancy that required or would require chemotherapy or radiation therapy within 1 year prior to randomization through the LFU Visit.
3. Patients with creatinine clearance (CrCl) of ≤30 mL/min, as estimated by the Cockcroft Gault formula, at Screening.
4. Patients with hemoglobin <10.0 g/dL or <6.2 mmol/L at Screening; donation of blood or plasma within 28 days prior to randomization; or symptomatic loss of blood or hemorrhage within 28 days prior to randomization.
5. Patients with severe hemoptysis within 28 days prior to randomization, defined as >100 mL over any 24-hour period or severe or extremely severe hemoptysis.
6. Patients with severe hepatic impairment, as evidenced by alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × upper limit of normal (ULN) or total bilirubin >2 × ULN, or clinical signs of cirrhosis or end-stage hepatic disease.
7. Patients who are pregnant or breastfeeding.
8. Patients with a mean QT interval corrected using Fridericia's formula (QTcF) >480 msec based on triplicate 12-lead ECGs at Screening.
9. Patients with an immunodeficiency or an immunocompromised condition and risk for an opportunistic pulmonary infection.
10. Patients with an anticipated start of new non-study antimycobacterial therapy to be administered at any time between Screening and Month 6.
11. Patients who have received any investigational medication during the 30 days or 5 half-lives, whichever is longer, prior to randomization.
12. Patients with any prior exposure to epetraborole.
13. Patients with any condition that, in the opinion of the Investigator, interferes with the ability to safely complete the study or adhere to study requirements, including the patient's inability or unwillingness to comply with all study assessments and visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Phase 2: Assessment of novel Patient Reported Outcome instrument psychometric properties | Screening (Day -14 to Day -7) to Month 6 + 1 week
  Assessment of novel Patient Report outcomes
Phase 2: Percentage of Participants Achieving Clinical Response | Baseline to Month 6
  Detection of within-patient changes in symptoms reported in a novel Patient-Reported Outcome (PRO) instrument at Month 3 and Month 6.
Phase 2: Adverse Event Profile of 500 mg Once Daily Dose of Epetraborole | Baseline to Month 16
  Percentage of Participants reporting treatment emergent adverse events
Phase 3: Percentage of Participants Achieving Clinical Response | Baseline to Month 6
  Detection of within-patient changes in symptoms reported in a novel Patient-Reported Outcome (PRO) instrument at Month 6

SECONDARY OUTCOMES:
Phase 2: Percentage of Participants Achieving Culture Conversion | Baseline to Month 6
  Sputum conversion will be assessed using culture conversion based on 3 consecutive monthly negative sputum cultures for MAC by Month 6.
Phase 2: Percentage of Participants Achieving Microbiological Improvement | Baseline to Month 6
  Microbiological improvement will be assessed at Month 3 and Month 6 using decrease in MAC colony counts of ≥1 category.
Phase 2: Change from Baseline in QOL-B Respiratory Domain PRO | Baseline to Month 6
  Mean change from baseline in Quality of Life - Bronchiectasis (QOL-B) respiratory domain score measured monthly through Month 6.
Phase 2: Change from Baseline in NTM Symptoms Module PRO | Baseline to Month 6
  Mean change from baseline in NTM Symptoms Module score measured monthly through Month 6.
Phase 2: Change from Baseline in SGRQ-C PRO | Baseline to Month 6
  Mean change from baseline in total Saint George's Respiratory Questionnaire for COPD Patients (SGRQ-C) score measured monthly through Month 6
Phase 2: Concordance Analysis of PRO-based Clinical Response and Microbiological Response | Baseline to Month 6
  Concordance between clinical response in a novel Patient-Reported Outcome (PRO) instrument and microbiological response will be assessed at Months 3 and 6. Microbiological response will be assessed using both sputum culture conversion and microbiological improvement.
Phase 2: Percentage of Participants with Reinfection | Baseline to Month 16
  By-subject reinfection will be assessed at Month 6, End of Therapy, and Late Follow-up. Reinfection is defined as a new pulmonary MAC infection caused by pathogen[s] different from the baseline MAC isolate.
Phase 2: Percentage of Participants with Relapse | Baseline to Month 16
  By-subject relapse will be assessed at Month 6, End of Therapy, and Late Follow-up. Relapse is defined as a pulmonary MAC infection caused by the same baseline MAC isolate after initial culture conversion.
Phase 2: Maximum plasma concentration (Cmax) of epetraborole | Day 1 and Day 29
  Cmax is the maximum plasma concentration of epetraborole estimated by population PK model.
14. Phase 2: Area Under the Plasma Concentration-Time Curve from Time Point 0 Hours Until 24 hours [AUC(0-24)] post dose | Day 29
  AUC(0-24) is defined as area under the plasma concentration-time curve of epetraborole from timepoint 0 hours until 24 hours post dose estimated by population PK model.
Phase 2: Volume of distribution (Vd) of epetraborole | Day 29
  Vd is the apparent volume of distribution of epetraborole estimated by population PK model.
Phase 3: Percentage of Participants Achieving Culture Conversion | Baseline to Month 6
  Sputum conversion will be assessed using culture conversion based on 3 consecutive monthly negative sputum cultures for MAC by Month 6.
Phase 3: Percentage of Participants Achieving Microbiological Improvement | Baseline to Month 6
  Microbiological improvement will be assessed at Month 3 and Month 6 using decrease in MAC colony counts of ≥1 category.
Phase 3: Change from Baseline in QOL-B Respiratory Domain PRO | Baseline to Month 6
  Mean change from baseline in Quality of Life - Bronchiectasis (QOL-B) respiratory domain score measured monthly through Month 6.
Phase 3: Change from Baseline in NTM Symptoms Module PRO | Baseline to Month 6
  Mean change from baseline in NTM Symptoms Module score measured monthly through Month 6.
Phase 3: Change from Baseline in SGRQ-C PRO | Baseline to Month 6
  Mean change from baseline in total Saint George's Respiratory Questionnaire for COPD Patients (SGRQ-C) score measured monthly through Month 6.
Phase 3: Concordance Analysis of PRO-based Clinical Response and Microbiological Response | Baseline to Month 6
  Concordance between clinical response in a novel Patient-Reported Outcome (PRO) instrument and microbiological response will be assessed at Months 3 and 6. Microbiological response will be assessed using both sputum culture conversion and microbiological improvement
Phase 3: Percentage of Participants with Reinfection | Baseline to Month 16
  By-subject reinfection will be assessed at Month 6, End of Therapy, and Late Follow-up. Reinfection is defined as a new pulmonary MAC infection caused by pathogen[s] different from the baseline MAC isolate.
Phase 3: Percentage of Participants with Relapse | Month 6, End of Therapy and Late Follow-up
  By-subject relapse will be assessed at Month 6, End of Therapy, and Late Follow-up. Relapse is defined as a pulmonary MAC infection caused by the same baseline MAC isolate after initial culture conversion.
Phase 3: Adverse Event Profile of 500 mg Once Daily Dose of Epetraborole | Baseline to Month 16
  Percentage of Participants reporting treatment emergent adverse events.
Phase 3: Maximum plasma concentration (Cmax) of epetraborole | Day 1 and Day 29
  Cmax is the maximum plasma concentration of epetraborole estimated by population PK model.
Phase 3: Area Under the Plasma Concentration-Time Curve from Time Point 0 Hours Until 24 hours [AUC(0-24)] post dose | Day 29
  AUC(0-24) is defined as area under the plasma concentration-time curve of epetraborole from timepoint 0 hours until 24 hours post dose estimated by population PK model.
Phase 3: Volume of distribution (Vd) of epetraborole | Day 29
  Vd is the apparent volume of distribution of epetraborole estimated by population PK model.

CONTACTS AND LOCATIONS:
Locations (91):
- United States (49):
  - 423032, Birmingham, Alabama
  - 423037, Tucson, Arizona
  - 423070, Sacramento, California
  - 423069, San Francisco, California
  - 423006, Stanford, California
  - 423068, Washington D.C., District of Columbia
  - 423075, Bay Pines, Florida
  - 423018, DeLand, Florida
  - 423034, Kissimmee, Florida
  - 423033, Tampa, Florida
  - 423054, Tampa, Florida
  - 423047, Tampa, Florida
  - 423038, Vero Beach, Florida
  - 423027, Atlanta, Georgia
  - 423076, Indianapolis, Indiana
  - 423029, Iowa City, Iowa
  - 423015, Kansas City, Kansas
  - 423063, Wichita, Kansas
  - 423065, Jefferson, Louisiana
  - 423042, New Orleans, Louisiana
  - 423060, Baltimore, Maryland
  - 423003, Baltimore, Maryland
  - 423074, Boston, Massachusetts
  - 423061, Boston, Massachusetts
  - 423078, Ann Arbor, Michigan
  - 423031, Rochester, Minnesota
  - 423008, St Louis, Missouri
  - 423004, Omaha, Nebraska
  - 423009, Lebanon, New Hampshire
  - 423024, Manhasset, New York
  - 423014, New York, New York
  - 423013, New York, New York
  - 423071, Chapel Hill, North Carolina
  - 423072, Charlotte, North Carolina
  - 423017, Durham, North Carolina
  - 423039, Winston-Salem, North Carolina
  - 423079, Cleveland, Ohio
  - 423082, Oklahoma City, Oklahoma
  - 423007, Portland, Oregon
  - 423002, Philadelphia, Pennsylvania
  - 423058, Philadelphia, Pennsylvania
  - 423045, Charleston, South Carolina
  - 423001, Charleston, South Carolina
  - 423067, Nashville, Tennessee
  - 423081, Fort Worth, Texas
  - 423005, Tyler, Texas
  - 423012, Charlottesville, Virginia
  - 423080, Edmonds, Washington
  - 423011, Milwaukee, Wisconsin
- Australia (7):
  - 501005, Concord, New South Wales
  - 501007, Birtinya, Queensland
  - 501003, Chermside West, Queensland
  - 501001, Greenslopes, Queensland
  - 501008, Perth, Western Australia
  - 501004, Clayton
  - 501002, South Brisbane
- Japan (29):
  - 215019, Aichi
  - 215026, Aomori
  - 215004, Fukuoka
  - 215025, Fukuoka
  - 215016, Fukuoka
  - 215006, Gifu
  - 215030, Hiroshima
  - 215014, Hokkaido
  - 215028, Ibaraki
  - 215018, Ishikawa
  - 215020, Ishikawa
  - 215017, Kanagawa
  - 215021, Kitakyushu
  - 215009, Kyoto
  - 215013, Kyoto
  - 215022, Mie
  - 215023, Nagano
  - 215002, Niigata
  - 215029, Osaka
  - 215008, Osaka
  - 215012, Osaka
  - 215001, Tokyo
  - 215005, Tokyo
  - 215024, Tokyo
  - 215003, Tokyo
  - 215027, Tokyo
  - 215010, Wakayama
  - 215007, Yamaguchi
  - 215011, Yokohama
- South Korea (6):
  - 219003, Gwangju
  - 219005, Incheon
  - 219001, Seongnam-si
  - 219002, Seoul
  - 219007, Seoul
  - 219008, Seoul